CLINICAL TRIAL: NCT02402153
Title: Evaluation of Hypo-Safe Hypoglycaemia Alarm Device - the Pilot 2 Study - Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNEEG Medical A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pilot 2_health_v2_August 27th
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Evaluation of subcutaneous EEG recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sydvestjysk Hospital (Other): Investigation of EEG recording with the Hyposafe device
  Interventions: Device: Hyposafe device

INTERVENTIONS:
Device: Hyposafe device — Subcutaneous EEG recorder for EEG measurements

SUMMARY:
The objective of this pilot trial is to demonstrate the safety and the performance of the Hyposafe hypoglycaemia alarm device before conducting clinical trials in type 1 diabetes patients.

DETAILED DESCRIPTION:
1. Safety: To evaluate safety issues related to implantation and use of the Hyposafe hypoglycaemia alarm device.
2. Performance: To evaluate the performance of the Hyposafe hypoglycaemia alarm device.
3. Usability: To obtain information about the subjects use and acceptance of the Hyposafe Hypoglycaemia alarm device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age 18-70 years
* For female participants: Not pregnant and, if child bearing potential, usage of reliable anti-contraceptive method during the study period

Exclusion Criteria:

* Severe cardiac disease

  * History of myocardial infarction
  * Cardiac arrhythmia
* Previous stroke or cerebral haemorrhage and any other structural cerebral disease
* Active cancer or cancer diagnosis within the past five years
* Uraemia defined as s-creatinine above 3 times upper reference value
* Liver disease defined as s-alanine aminotransferase (s-ALAT) above 3 times upper reference interval
* Epilepsy
* Use of antiepileptic drugs for any purposes
* Clinical important hearing impairment
* Use of active implantable medical device including

  * Pacemaker and Implantable Cardioverter Defibrillator (ICD-unit)
  * Cochlear implant
* Use of following drugs

  * Chemotherapeutic drugs of any kind
  * Methotrexate
  * Third generation antipsychotic drugs (aripiprazole, quetiapine, clozapine, ziprasidone, paliperidone, risperidone, sertindole, amisulpride, olanzapine)
* Abuse of alcohol (defined as consumption of > 250g alcohol (in Danish: 21 "genstande")) per week or abuse of any other neuro-active substances
* Infection at the site of device-implantation
* Any haemorrhagic disease
* Diving (snorkel diving allowed) or parachute jumping
* Patients that are judged incapable to understand the patient information or who are unlikely to complete the investigation for any reason
* Persons operating MRI scanners.
* Persons operating handheld transceivers for communication (e.g. within the police, medical, fire, air traffic control, marine or military).
* Persons working at broadcast stations for television or FM/DAB radio.
* Persons performing extreme sport.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birger Thorsteinsson, MD, DMSc, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Sydvestjysk Hospital, Esbjerg, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Sydvestjysk Hospital: Observational EEG recording with the Hyposafe device
  Hyposafe device: Subcutaneous EEG recorder for EEG measurements
Period: Overall Study
Arm/Group | Sydvestjysk Hospital
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sydvestjysk Hospital
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 37 [25 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 18
Weight [Mean (Full Range); unit: Kg] | 87 [63 to 126.3]
Height [Mean (Full Range); unit: Centimeter] | 175.7 [153.5 to 205]
Blood pressure (systolic) [Mean (Full Range); unit: mmHg] | 123 [105 to 168]
Blood pressure (diastolic) [Mean (Full Range); unit: mmHg] | 79 [65 to 102]

OUTCOME MEASURES:

1. Primary Outcome: Performance: EEG Recordings - Impedance
Description: The EEG performance was measured as the mean impedance as a function of time. An impedance value below 5 kOhm is considered very good.
Time Frame: 1 month
Population: Exclusion of data points (n=6) in the analysis:
  A software bug resulted in no data storage (n=2). After a protocol amendment, EEG data was collected for the first 3 weeks only. The subsequent 2 weeks subjects were monitored, but EEG data not collected (n=4).
Measure: Mean (Standard Deviation); unit: Impedance (kOhm)
Arm/Group | Sydvestjysk Hospital
Number analyzed (Participants) | 12
Impedance (kOhm) | 2.3 (0.13)

2. Primary Outcome: Performance: EEG Quality
Description: The power spectrum densities from the two modalities were directly compared on an integer scale from -5 to 5, where "-5" signifies that the scalp EEG was of much higher quality than the subcutaneous. "0" means they were of equal quality and "5" means the subcutaneous signal was of much higher quality
Time Frame: 1 month
Population: Exclusion of data points (n=5) in the analysis: A software bug and usage error of the control setup.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Sydvestjysk Hospital
Number analyzed (Participants) | 13
Score | 0.4 (0.8)

3. Primary Outcome: Performance: Continuous EEG
Description: Average time of EEG recordings (hours/day)
Time Frame: 1 month
Population: Exclusion of data points (n=8) in the analysis:
  A software bug resulted in reduced data storage (n=4). After an amendment to the study protocol, EEG data was collected for the first 3 weeks. The subsequent 2 weeks subjects were monitored, but EEG data not collected (n=4).
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Sydvestjysk Hospital
Number analyzed (Participants) | 10
hours/day | 20.3 (2.1)

4. Secondary Outcome: Usability: Reported Discomfort During Day While Wearing the Device
Description: The discomfort during the day was recorded by the study subject every day wearing the device. Reported discomfort was evaluated by the following question: "How much do you agree with the following statement: There has been no discomfort while wearing the HypoSafe device during day?". The scale ranged from 1 to 5 (strongly agree = 5, agree = 4, neutral = 3, disagree = 2, strongly disagree=1).
Time Frame: 1 month
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Sydvestjysk Hospital
Number analyzed (Participants) | 18
units on a scale | 4.1 [2.5 to 5]

5. Secondary Outcome: Usability: Reported Discomfort During Night While Wearing the Device
Description: The discomfort during the night was recorded by the study subject every night wearing the device. Reported discomfort was evaluated by the following question: "How much do you agree with the following statement: There has been no discomfort while wearing the HypoSafe device during night?". The scale ranged from 1 to 5 (strongly agree = 5, agree = 4, neutral = 3, disagree = 2, strongly disagree=1).
Time Frame: 1 month
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Sydvestjysk Hospital
Number analyzed (Participants) | 18
units on a scale | 3.8 [1.75 to 5]

6. Secondary Outcome: Usability: Reported Discomfort Related to the Implant in the Beginning of the Study
Description: The discomfort was recorded by the study subjects 19±4 days after implantation. Reported discomfort was evaluated by the following question: "How much do you agree with the following statement: I have not experienced any implant discomfort the past two days?". The scale ranged from 1 to 5 (strongly agree = 5, agree = 4, neutral = 3, disagree = 2, strongly disagree=1).
Time Frame: 19±4 days after implantation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sydvestjysk Hospital
Number analyzed (Participants) | 18
units on a scale | 3.8 (1.3)

7. Secondary Outcome: Usability: Reported Discomfort Related to the Implant at the End of the Study
Description: The discomfort was recorded by the study subjects 51±3 days after implantation. Reported discomfort was evaluated by the following question: "How much do you agree with the following statement: I have not experienced any implant discomfort the past two days?". The scale ranged from 1 to 5 (strongly agree = 5, agree = 4, neutral = 3, disagree = 2, strongly disagree=1).
Time Frame: 51±3 days after implantation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sydvestjysk Hospital
Number analyzed (Participants) | 18
units on a scale | 4.3 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first subject first visit to last subject last follow-up. Total period for AE collection was 2 years.
Description: Adverse Events (AEs) were collected as defined in the International Standards Organizations (ISO): ISO 14155 Clinical investigation of medical devices for human subjects - Good clinical practice. All AEs were reported regardless of being related or unrelated to the device
Arm/Group | Sydvestjysk Hospital
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 15/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sydvestjysk Hospital (N=18)
Ventricular extrasystoles (Cardiac disorders) | 1 — Not device related
Includes either ear swelling, ear discomfort, ear pain, or ear deformity acquired (Ear and labyrinth disorders) | 7 — Device related
Vomiting and diarrhoea (Gastrointestinal disorders) | 1 — Not device related
Includes either implant site haematoma, discomfort or implant site pain (General disorders) | 3 — Device related
Includes either nasopharyngitis, ear infection or food poisoning (Infections and infestations) | 6 — Not device related
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Not device related
Includes either headache, post procedural headache or migrane (Nervous system disorders) | 4 — Device related
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 — Not device related
Hypertension (Vascular disorders) | 1 — Not device related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data is the property of UNEEG medical A/S. The PI is offered co-authorship for publications related to the investigation. If the PI does not agree on the interpretation of the results, then the PI have the right to publish and present the results.